CLINICAL TRIAL: NCT03933358
Title: Effect of Thyroid Hormone on Post-Myocardial Infarction Remodeling and Prognosis in STEMI Patients
Acronym: ThyREST
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Principal Investigator, Hongwei Li, MD, Prof., Beijing Friendship Hospital
Other Study IDs: BFH-Thyroid and STEMI
Record Dates: First submitted 2019-04-29; First posted 2019-05-01 (Actual); Last update posted 2019-05-03 (Actual); Status verified 2019-05

CONDITIONS: Thyroid; Cardiac Remodeling, Ventricular; STEMI
MeSH Terms: conditions — Thyroid Diseases; Ventricular Remodeling; ST Elevation Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Euthyroid
  Interventions: Other: Thyroid hormone levels
- Low T3: low triiodothyronine syndrome
  Interventions: Other: Thyroid hormone levels

INTERVENTIONS:
Other: Thyroid hormone levels — This is an observational study. Exposure: Different thyroid hormone levels.

SUMMARY:
This study aims to determine whether thyroid hormone levels are predictive of cardiac remodeling following myocardial infarction and the prognosis in patients with STEMI receiving primary percutaneous coronary intervention.

ELIGIBILITY:
Inclusion Criteria:

* with a confirmed STEMI diagnosis
* undergoing primary percutaneous coronary intervention (presenting <12h after symptom onset)
* patients agreed and provided informed consent

Exclusion Criteria:

* past history of myocardial infarction or percutaneous coronary intervention or coronary artery bypass graft
* past history of heart failure (LVEF<40%) or myocardiopathy or atrial fibrillation
* past history of thyroid diseases, or were treated with amiodarone, dopamine, or corticosteroids before hospital admission
* contraindicating to cardiac magnetic resonance imaging

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients admitted to Beijing Friendship Hospital with a confirmed STEMI diagnosis undergoing primary percutaneous coronary intervention
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2019-05-01 (Estimated); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
MACE (major adverse cardiovascular events) | 12 months
  cardiovascular death, re-infarction, revascularization, and stroke

SECONDARY OUTCOMES:
adverse cardiac remodeling | 6 months
  a cut-off value of 12% change in left ventricular end-diastolic volume between the acute and follow-up magnetic resonance scans
all-cause death | 12 months
  death caused by all reason

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Friendship Hospital, Capital Medical University, Beijing, China